CLINICAL TRIAL: NCT04807946
Title: A Prospective Observational Study on the Variables Affecting the Risk of Inferior Alveolar Nerve Damage During Lower Third Molar Surgery With Nerve/Root Proximity
Brief Title: Study on the Risk of Inferior Alveolar Nerve Damage During Lower Third Molar Surgery
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Pippi Roberto, Professor, University of Roma La Sapienza
Other Study IDs: 4111
Record Dates: First submitted 2021-03-03; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Mandibular Nerve Injury
MeSH Terms: conditions — Mandibular Nerve Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: lower third molar extraction — All surgeries were performed by the same expert surgeon (RP), with the buccal approach using local anesthesia, and included the following maneuvers:
  * luxation of the coronal portion of the tooth/root in an ipsilateral or parallel direction with respect to the IAN position and running, in order to minimize nerve compression;
  * post-extraction residual bone cavity inspection using a Zeiss 4x300 magnification optical system to better identify intra-operative nerve exposure.
  No material was inserted into the residual cavity, neither by regeneration nor by haemostasis.
  After one week, sensitivity was tested on both sides with the tactile test using a 27-gauge needle tip and, if a difference was found, the patient was followed up once a week for the first month and every two weeks thereafter, until he/she reported to perceive the pin-prick test in the affected side the same way as the healthy side.

SUMMARY:
Objective The present study aimed to evaluate which factors were statistically associated with a greater probability of inferior alveolar nerve (IAN) damage during lower third molar surgery.

Study Design A prospective observational study was performed at the Oral Surgery Unit of the Umberto I Hospital on 92 patients which underwent surgical extraction of a lower third molar, that was radiographically overlapped to the mandibular canal. All surgeries were performed by the same expert surgeon. A principal component analysis and the exact two-tailed Fisher test were used.

DETAILED DESCRIPTION:
Exclusion criteria were the following:

* lower third molar buds;
* lack of contiguous second molar;
* wide cyst-like areas or severe osteo-metabolic/tumor pathologies associated with the lower third molar;
* pre-operative neurosensory deficit related to IAN on the side where surgery was to be performed.

Clinical and radiographic data were noted on a special chart, developed in four areas concerning the patient's personal data, pre-operative case evaluation, surgical technique, and post-operative course.

Assessment of surgical difficulty was reached using a modified Pederson's scale by assigning a 1 to 3 score to each of the following variables: tooth inclination (mesioangular/vertical = 1; horizontal = 2; distoangular = 3), depth of impaction (modified Winter classification: A/B = 1; C1 = 2; C 2= 3), Pell & Gregory class (I = 1; II = 2; III = 3), root morphology (fused or slightly divergent = 1; strongly divergent = 2; presence of apical anomalies = 3), proximity to the IAN (none = 1; contiguity = 2; embrication = 3) and maximum mouth opening (> 4 cm = 1; 3-4 cm = 2; < 3 cm = 3). For each extracted third molar, a total score between 6 and 18 was therefore obtained.

All surgeries were performed by the same expert surgeon (RP), with the buccal approach using local anesthesia, and included the following maneuvers:

* luxation of the coronal portion of the tooth/root in an ipsilateral or parallel direction with respect to the IAN position and running, in order to minimize nerve compression;
* post-extraction residual bone cavity inspection using a Zeiss 4x300 magnification optical system to better identify intra-operative nerve exposure.

No material was inserted into the residual cavity, neither by regeneration nor by haemostasis.

After one week, sensitivity was tested on both sides with the tactile test using a 27-gauge needle tip and, if a difference was found, the patient was followed up once a week for the first month and every two weeks thereafter, until he/she reported to perceive the pin-prick test in the affected side the same way as the healthy side.

ELIGIBILITY:
Inclusion Criteria:

* orthopantomographic superimposition between the lower third molar and at least the upper half of the mandibular canal, associated or not with the presence of one or more radiographic signs of proximity among those proposed by Rood and Shehab (1990):
* 3-dimensional radiographic examination with a CT software;
* any type of lower third molar impaction.

Exclusion Criteria:

* lower third molar buds;
* lack of contiguous second molar;
* wide cyst-like areas or severe osteo-metabolic/tumor pathologies associated with the lower third molar;
* pre-operative neurosensory deficit related to IAN on the side where surgery was to be performed.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Each patient came to the Oral Surgery Unit of the Umberto I Hospital, Department of Odontostomatological and Maxillofacial Sciences, Sapienza University of Rome to extract the lower third molar that present the inclusion criteria. Patients were enrolled only after giving consent to participate in the study. Consent to statistical treatment of clinical and radiographic data was also obtained from all patients.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-02-08 (Actual)

PRIMARY OUTCOMES:
Assessment of sensitivity alteration after extraction | After 7 days, at the suture removal, the sensitivity was tested.
  sensitivity in the territory of innervation of the inferior alveolar nerve, sensitivity was tested on both sides with the tactile test using a 27-gauge needle tip and, if a difference was found, the patient was followed up once a week for the first month and every two weeks thereafter, until he/she reported to perceive the pin-prick test in the affected side the same way as the healthy side.
Change of Sensitivity after every week for the first month | in case of alteration the checks were carried out every weeks up to 30 days
  sensitivity in the territory of innervation of the inferior alveolar nerve, sensitivity was tested on both sides with the tactile test using a 27-gauge needle tip and, if a difference was found, the patient was followed up once a week for the first month and every two weeks thereafter, until he/she reported to perceive the pin-prick test in the affected side the same way as the healthy side.
Change of Sensitivity after every two week for the second month until resolution | in case of alteration over 30 days we checks every 2 weeks until resolution, up to 365 days.
  sensitivity in the territory of innervation of the inferior alveolar nerve, sensitivity was tested on both sides with the tactile test using a 27-gauge needle tip and, if a difference was found, the patient was followed up once a week for the first month and every two weeks thereafter, until he/she reported to perceive the pin-prick test in the affected side the same way as the healthy side.